CLINICAL TRIAL: NCT05530148
Title: Investigating the Effects of a Complex, Partnered Martial Arts-based Intervention on Processing Speed in Comparison to Less Complex Exercise in Low-active Adults.
Brief Title: Effects of a Complex, Partnered Martial Arts-based Intervention on Cognitive Processing.
Acronym: MATRICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23222
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Change; Processing, Visual Spatial
Keywords: Cognitive Performance; Complex movement; Skill Acquisition; Processing Speed
MeSH Terms: conditions — Spatial Processing

STUDY DESIGN:
Intervention Model Description: The study is a single-blind randomized trial with parallel groups design involving an experimental exercise and an exercise comparison.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to group allocation. Participants will not be masked from knowledge of the other group, but will only receive the training from one specific training group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Martial Arts Group (Experimental): Participants will be trained in the martial arts exercises using both in-person group sessions and asynchronous remote learning via video content distributed to them each week. Participants will be asked to attend as many of the 24 in-person sessions as they can. Heartrate will be monitored periodically to make sure the intensity of exercise is consistent with mild to moderate cardiovascular exercise as in the active comparator.
  Interventions: Behavioral: Martial Arts Training Group
- Flexing, Toning and Balance (Active Comparator): Flexibility, Toning and Balance or FTB will be used to refer to our resistive exercise comparison. As in the experimental group, participants will be asked to attend as many of the 24 in-person intervention sessions as they can, whilst also practicing the exercises remotely via video content distributed to them. The remote portion of this intervention will be asynchronous. Heart-rate will be monitored periodically to make sure the intensity of exercise is consistent with mild to moderate cardiovascular exercise as in the martial arts experimental group.
  Interventions: Behavioral: Flexing, Toning and Balance

INTERVENTIONS:
Behavioral: Martial Arts Training Group — Participants in the experimental intervention group will attend as many of the 24 in-person training sessions as possible, and complete remote solo training at their leisure, for the duration of the intervention period. During the in-person sessions, they will be instructed in the three exercises practiced in the experimental group, known as hubud, chi sau and padwork. Hubud is a turn-based, partnered, coordination drill involving moves derived from numerous martial arts, most often seen in the Filipino martial art of Kali. Chi Sau is a simultaneous contact drill from Chinese Kung Fu, specifically the Wing Chun school. Padwork is an amalgam of punching and kicking combinations used against focus pads or padded sticks to improve coordination, most commonly seen in kickboxing and Muay Thai. Participants will aim to reach a level of comfort and competency in the basic, non-competitive aspects of these exercises by the end of their participation in this intervention.
  Arms: Martial Arts Group
Behavioral: Flexing, Toning and Balance — Participants in the active comparator group will attend as many of the 24 in-person training sessions as possible, and complete remote solo training at their leisure, for the duration of the intervention period. During the in-person sessions, participants will start with a 5-minute warmup of basic joint mobilization exercises and dynamic stretching techniques. After this, participants will engage in a mild intensity circuit of exercises using resistance bands, bodyweight exercises and stability/balance exercises for approximately 50 minutes. The last 5 minutes of the session will be left for cooldown exercises and light stretching. Heartrate will be monitored regularly in order to prevent these exercises exceeding the relative intensity of the Martial Arts intervention group. Participants will be allowed to talk and interact with research assistants in order to keep socialization effects consistent across groups.
  Other Names: Resistive Exercise Group; Active Comparison Group
  Arms: Flexing, Toning and Balance

SUMMARY:
The investigators' study is designed to test whether prolonged exposure to a martial arts-based intervention (three complex, partner exercises based on Filipino, Chinese and Thai martial arts practices), can improve cognitive processing to a greater degree than resistive exercise of a similar intensity.

DETAILED DESCRIPTION:
This two-group randomized controlled trial will compare the effects of a martial arts intervention vs. resistive exercise condition. The martial arts intervention will consist of partnered, coordinated exercises drawn from south-east Asian martial arts, including Fillipino Kali, Chinese Wing Chun Kung Fu and Muay Thai (also known as Thai Boxing). Participants will be trained in the fundamental movements of the exercises known as hubud, chi sau and padwork. Participants will also have the history, cultural significance, risks and purpose of these exercises explained to them throughout the study.

The resistive exercise comparator group will use a series of bodyweight resistance, band resistance and postural exercises to match the duration and exercise intensity of the martial arts intervention group, under the supervision of trained research assistants. Participants will also receive information on aerobic exercise and the Physical Activity Guidelines for Americans 2020.

All participants, regardless of group, will be assessed for martial arts and exercise experience once at baseline.

All participants will be tested for cognitive performance change. Baseline and follow-up computerized cognitive testing will take place at a specified testing facility and psychosocial questionnaires will be delivered remotely via a Qualtrics-powered survey. After baseline testing, participants will be asked to attend as many sessions (maximum 24 sessions) delivered over the course of an 8-week intervention period as they can, approximately 1 hour each. Follow-up testing will be administered more than 48 hours post-intervention to minimize established acute adaptive responses to exercise.

The investigators hypothesize the martial arts training intervention group will exhibit a greater increase in performance of cognitive processing tasks when compared to less complex movement patterns involved in the resistive exercise group.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between the ages of 18-45 years reporting lower levels of physical activity (sedentary or mild physical activity levels only)

Exclusion Criteria:

* Anyone who is physically active (≥30 minutes, 3 or more times/week, for the last 3 months) and/or a regular practitioner of martial arts and/or highly complex coordination drills such as dance and exercises related to coordinated movement (≥30 minutes, 3 or more times/week, for the last 3 months).
* Anyone with serious chronic medical conditions that would preclude them from participating without a physician present, or anyone with a risk of seizure, or anyone having psychiatric and/or neurological disorders.
* Pregnant women or anyone with recent (within the two months) surgery on their shoulders, elbows, knees or hips.
* Anyone who is currently diagnosed with depression and is receiving treatment (medication or counselling) for their depression.
* Anyone incapable of performing the following movements at a moderate intensity- sitting, standing, kicking, pulling, pushing, bending one's elbows or bending one's knees.
* Anyone who scores 1 or more on the Physical Activity Readiness Questionnaire
* Anyone refusing or unwilling to be randomized into either of the conditions.
* Anyone with insufficient proficiency (fluency) in English to understand the
* Anyone with blood pressure readings exceeding our safety limits (systolic >160 and diastolic >90)
* Anyone who has tested positive for COVID-19 within the last 60 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Processing Speed (Latent Factor) | 8 weeks
  Cognitive processing speed will be modeled within a latent variable framework reflecting standardized scores from four heterogeneous assessments involving visual stimuli. Performance for all of these tasks will be measured by number of correct responses (accuracy) as well as reaction/decision-making times.

SECONDARY OUTCOMES:
Godin Leisure-Time Exercise Questionnaire | 8 weeks
  This is a 4-item assessment of physical activity. Respondents are asked the frequency they engage in strenuous, moderate and mild activity for 15 minutes or more as part of their free time. Weekly leisure time exercise is measured using a weighted formula as follows:
  (9 x strenuous PA) + (5 x moderate PA) + (3 x light PA)
Memory | 8 weeks
  Frequency of Forgetting is a 10-item scale asking participants to score on a 1-10 Likert scale how often they forget or have difficulty remembering certain things. On this scale, 1 = Always and 10 = Never. The measure is typically scored as a sum of all responses, with a higher number indicating better memory/recall and lower numbers indicating poorer memory/recall. The first item also serves as a standalone measure.
Enjoyment of Exercise | 8 weeks
  The Physical Activity Enjoyment Scale (PACES) was originally an 18-item scale for assessing PA enjoyment, and has been further refined and psychometrically tested by Mullen and his colleagues (Massey et al 2021; Mullen et al 2011). The 7-item version is a reliable and time-invariant measure. The scale asks participants "How do you feel at the moment about the physical activity you have been doing?" and responses are provided on 7-point Likert scales. For example, "Its no fun at all" and "Its a lot of fun" represent bipolar anchors. Items are added and averaged whereby higher scores reflect greater levels of enjoyment.
Perceived Mental Fatigue | 8 weeks
  A novel, 7-item assessment of current state of mental fatigue will be used (example items include "My thoughts easily wander," "My thinking requires effort.") The scales response ranges from 1 (not true at all) to 5 (very true) and all items are summed and averaged whereby higher scores indicated greater mental fatigue.
Perceptions of Mastery | 8 weeks
  Perceptions of Mastery has four items scored on a 5-point likert scale. Two items ask participants to rate their current level of knowledge/mastery and two items address performance and skill status; with -2 meaning 'rapidly declining' and +2 meaning 'rapidly improving.' Scores are summed and then average to give a measure of perceived mastery.

OTHER OUTCOMES:
Grip strength task | 8 weeks
  A dynamometer will be used to assess grip strength. Under supervision, participants will engage in two trials per hand (unless each trial results in an increasing or identical score, at which point a third trial will be used). The highest score, as well as an average of the two highest scores, will be recorded as measures of grip strength from this task.
Dot task | 8 weeks
  Agility will be assessed with a timed, choreographed sequence of steps on a dotted floor mat (positioned in an X-pattern). Performance will be based on how quickly (measured in seconds) they can perform the prescribed, choreographed sequence.
Trail-Making Test | 8 weeks
  The trail-making test is a global cognition and spatial awareness assessment involving two parts. Respondents must complete each part as quickly as possible using a single, continuous pencil-drawn line. For Trails part A, the numbers 1-26 are randomly arranged on a sheet of paper and respondents are required to connect the numbers, in order, using a single pencil line. The pencil is not allowed to leave the paper until the task is complete. The same is true for Trails part B, but the sequence is now numero-alphabetic (1, A, 2, B, 3, C and so on). The task is complete when the participant reaches the end of the sequence. Performance will be measured by how long it takes the participant to complete parts A and B. Trails part B is considered the most challenging task and B-A is used as measure of executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Exercise, Technology, and Cognition Laboratory - Louise Freer Hall 284, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to the Primary investigator and Lead research assistant of this study.